CLINICAL TRIAL: NCT04696341
Title: The Effectiveness of a Novel Massage Method Matrix Rhythm Therapy in Chronic Neck Pain
Brief Title: The Effect of Matrix Rhythm Therapy in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Nur OYMAK SOYSAL, Lecturar, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25.01.2011/02
Record Dates: First submitted 2021-01-01; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain; Physical Disability
Keywords: Matrix Rhythm Therapy; Massage; Physical Therapy; Neck Pain
MeSH Terms: conditions — Chronic Pain; Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: All assessments were done by the same physiotherapist (FU) before therapy and at the end of treatment sessions. The physiotherapist who did the assessments did not know to which group the subjects were belonged. Another physiotherapist who was not informed about the results of the evaluation treated the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matrix Rhythm Therapy (Experimental): Group I (15 subjects) received 10 sessions as 5 sessions a week. Hot pack to cervical and upper thoracic regions, conventional TENS, therapeutic ultrasound, conventional massage and Matrix Rhythm Therapy were applied. Home-based exercise program and recommendations were also given to patients.
  Interventions: Procedure: Matrix Rhythm Therapy
- Control (Experimental): Group II (15 subjects) received 10 sessions as 5 sessions a week. Hot pack to cervical and upper thoracic regions, conventional TENS, therapeutic ultrasound and conventional massage were applied. Home-based exercise program and recommendations were also given to patients.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Matrix Rhythm Therapy — Hot pack to cervical and upper thoracic regions (20 min), conventional TENS (100 Hz for 40 μsec), therapeutic ultrasound (1 MHz for 5 min) and conventional massage (using stroking, kneading and friction techniques for 5 minutes) were applied as passive physiotherapy modalities. Normal range of motion exercises, posture exercises, stretching exercises and isometric exercises were instructed as part of active physiotherapy.Five sessions of MRT (2., 5., 6., 8., 10. sessions of combined physiotherapy programme) was added at combined physiotherapy to Matrix Rhythm Group. Matrix Rhythm Therapy was applied to cervical and thoracic regions using 10 Hz frequency for 30 min (15 min for right and left sides each) according to the instructions of the technique developer.
  Arms: Matrix Rhythm Therapy
Procedure: Control — Hot pack to cervical and upper thoracic regions (20 min), conventional TENS (100 Hz for 40 μsec), therapeutic ultrasound (1 MHz for 5 min) and conventional massage (using stroking, kneading and friction techniques for 5 minutes) were applied as passive physiotherapy modalities. Normal range of motion exercises, posture exercises, stretching exercises and isometric exercises were instructed as part of active physiotherapy.
  Arms: Control

SUMMARY:
Thirty individuals with chronic neck pain randomised into two groups. Group I (15 subjects) received a total of 10 sessions as 5 sessions a week.Hot pack to cervical and upper thoracic regions (20 minutes), conventional Transcutaneous Electrical Nerve Stimulation (TENS) (100 Hz for 40 μsec), therapeutic ultrasound (1 Megahertz (MHz) for 5 minutes) and conventional massage were applied. Five sessions of Matrix Rhythm Therapy (2., 5., 6., 8., 10. sessions of combined physiotherapy programme) was added at combined physiotherapy Group II. Matrix Rhythm Therapy was applied to cervical and thoracic regions using 10 Hz frequency for 30 minutes.

Pain intensity was measured using by a Visual Analogue Scale (VAS) measuring 10 cm. Muscle spasm in cervical region was assessed by using a VAS measuring 10 cm. Turkish version of Neck Disability Index (NDI) was used to assess the disability caused by neck pain. Turkish version of Beck Depression Inventory was used to assess emotional status of participants.

DETAILED DESCRIPTION:
The study included patients aged between 25-65 years who had neck pain for at least 3 months. Patients with radiculopathy who had motor findings, who underwent any operations due to neck problems, who had systemic, neurologic and psychiatric diseases, inflammatory or infectious diseases, history of malignity, congenital anomalies, who benefited from another therapy modality and the ones in whom physical therapy modalities could not be used due to contraindications (individuals with sensory disorders, who use cardiac pace maker) were excluded from the study.

A total of 36 individuals were randomly assigned into 2 groups. Randomization was allocated by numbered envelopes method. A total of 30 subjects (15 in Matrix Rhythm Therapy (MRT) group and 15 in CG) with neck pain due to mechanic causes like cervical discopathy, cervical arthrosis or myofascial pain syndrome were participated in this study.

All assessments were done by the same physiotherapist (FU) before therapy and at the end of treatment sessions. The physiotherapist who did the assessments did not know to which group the subjects were belonged. Another physiotherapist who was not informed about the results of the evaluation treated the patients.

Home-based exercise programs and recommendations were also given to patients. Matrix Rhythm Therapy is developed by Dr. Ulrich G. Randall at the university of Erlangen/Nuremberg. Longitudinal stroking, compression and spooning techniques are specific methods of MRT. Therapies of the patients were done by the physiotherapist who had certificate of MRT application.

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain for at least 3 months

Exclusion Criteria:

* radiculopathy with motor findings
* undergoing surgical operation for neck pathologies
* having a systemic , neurologic, psychiatric diseases
* inflammatory or infectious diseases targeting this region
* physical therapy modalities could not be used due to contraindications (individuals with sensory disorders, who use cardiac pace maker)
* pregnancy
* malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-25 (Actual); Primary Completion 2011-04-08 (Actual); Study Completion 2011-05-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Pain intensity was measured using by a Visual Analogue Scale (VAS) measuring 10 cm (0: I have no pain, 10: I have an intolerable pain). Higher scores mean a worse outcome.
Muscle spasm | Baseline
  Muscle spasm in cervical region was assessed by using a VAS measuring 10 cm (0: no spasm, 10: the most severe spasm). Higher scores mean a worse outcome.
Disability | Baseline
  Turkish version of Neck Disability Index (NDI) was used to assess the disability caused by neck pain. NDI is composed of a total of 10 questions of which 4 about subjective symptoms Each section is scored between 0 and 5. For total scores 0-4 no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, 35-50 complete disability
Emotional status | Baseline
  Turkish version of Beck Depression Inventory was used to assess emotional status of participants. Each question of the questionnaire which is composed of 21 questions is scored between 0 and 3. Higher scores than 17 mean risc for depression.

SECONDARY OUTCOMES:
Pain intensity | 2 weeks
  Pain intensity was measured using by a Visual Analogue Scale (VAS) measuring 10 cm
Muscle spasm | 2 weeks
  Muscle spasm in cervical region was assessed by using a VAS measuring 10 cm (0: no spasm, 10: the most severe spasm)
Disability | 2 weeks
  Turkish version of Neck Disability Index (NDI) was used to assess the disability caused by neck pain. NDI is composed of a total of 10 questions of which 4 about subjective symptoms Each section is scored between 0 and 5 caused by neck pain. For total scores 0-4 no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, 35-50 complete disability
Emotional status | 2 weeks
  Turkish version of Beck Depression Inventory was used to assess emotional status of participants. Each question of the questionnaire which is composed of 21 questions is scored between 0 and 3. Higher scores than 17 means risc for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Emine ASLAN TELCİ, Professor, Study Chair — Pamukkale University; Erhan ÖZFİDAN, Dr, Study Chair — Private Denizli Tekden Hospital
Locations (1):
- Sarayköy Vocational School, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because there is no web site to share my data

REFERENCES:
- [Result] Taspinar F, Aslan UB, Sabir N, Cavlak U. Implementation of matrix rhythm therapy and conventional massage in young females and comparison of their acute effects on circulation. J Altern Complement Med. 2013 Oct;19(10):826-32. doi: 10.1089/acm.2012.0932. Epub 2013 Apr 26. PMID 23621388
- [Result] Smidt N, de Vet HC, Bouter LM, Dekker J, Arendzen JH, de Bie RA, Bierma-Zeinstra SM, Helders PJ, Keus SH, Kwakkel G, Lenssen T, Oostendorp RA, Ostelo RW, Reijman M, Terwee CB, Theunissen C, Thomas S, van Baar ME, van 't Hul A, van Peppen RP, Verhagen A, van der Windt DA; Exercise Therapy Group. Effectiveness of exercise therapy: a best-evidence summary of systematic reviews. Aust J Physiother. 2005;51(2):71-85. doi: 10.1016/s0004-9514(05)70036-2. PMID 15924510
- [Result] Ylinen J. Physical exercises and functional rehabilitation for the management of chronic neck pain. Eura Medicophys. 2007 Mar;43(1):119-32. PMID 17369784